CLINICAL TRIAL: NCT03154554
Title: Epidemiology of Patients Consulting for Original LBP Spinal Adult Emergency Hautepierre and 3 Months Course of Care
Brief Title: Epidemiology of Patients Consulting for Original LBP Spinal Adult Emergency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6482
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Lumbar Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lumbar pain is an extremely common complaint in general population. The direct and indirect costs incurred in are a real public health problem.

Cohort studies show that improving symptoms after consultation for lumbar pain is insufficient, but there are few data on emergency medical and surgical services in France. In order to reflect on areas for improvement the investigators to carry out an inventory of consultations for lumbar pain emergencies of Hautepierre Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to adult emergencies in Hautepierre for lumbago pain, with or without sciatica,
* Age greater than or equal to 18 years
* Having signed non-opposition to participation in the study
* Having completed the initial questionnaire

Exclusion criteria:

* Spinal trauma in the month before the consultation
* Pain of non-spinal origin (pyelonephritis, colic Nephritic, aortic dissection ...)
* Non-Francophone Patients
* Patient under tutorship or under curatorship
* Patient under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to adult emergencies in Hautepierre for lumbago pain, with or without sciatica,
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
current clinical condition, lumbar antecedent and patient care questionnaires | At the time of consultation in the adult emergency department, 3 months after consultation in the adult emergency department
  The initial questionnaire focuses on the current clinical condition of the patient and his or her lumbar antecedent.
  The 3-month follow-up questionnaire focuses on the patient care during this period.

IPD SHARING:
Plan to Share IPD: No